CLINICAL TRIAL: NCT06950164
Title: Dynamic Changes of Ductus Arteriosus in < 31 Weeks Preterm Infants: an Observational Study
Acronym: PDA
Status: Active, not recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Chongqing Medical Center for Women and Children (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Chongqing Medical Center for Women and Children
Other Study IDs: ductus arteriosus
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Preterm; Ductus Arteriosus
Keywords: preterm; patent ductus arteriosus
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- observation group: in the group, no intervention was given, and the preterm infants were diagnosed with respiratory distress syndrome(RDS)
  Interventions: Other: observation group
- control group: in the group, no intervention was given, but the preterm infants were diagnosed without respiratory distress syndrome(RDS)
  Interventions: Other: control group

INTERVENTIONS:
Other: observation group — in the group, no intervention was given, and the preterm infants were diagnosed with respiratory distress syndrome(RDS)
  Groups: observation group
Other: control group — in the group, no intervention was given, but the preterm infants were diagnosed without respiratory distress syndrome(RDS)
  Groups: control group

SUMMARY:
The ductus arteriosus quickly closes itself. is an important channel connecting the maternal fetal circulation before birth. After birth, this ductus arteriosus generally no longer has a physical function, so ductus arteriosus quickly closes itself. The persistent presence of ductus arteriosus leads to significant pressure changes in the systemic and pulmonary circulation, which have adverse effects on extremely/very premature infants. Therefore, persistent patent ductus arteriosus (PDA) is a systemic disease.

DETAILED DESCRIPTION:
hemodynamic significant PDA(hsPDA) is a risk factor for intraventricular hemorrhage(IVH), bronchopulmonary dysplasia(BPD), necrotizing enterocolitis(NEC). A meta-analysis from Cochrane shows that compared to conservative treatment, drug therapy for PDA within 3 and 7 days after birth does not promote PDA closure and reduce the incidence of BPD. Therefore, there is currently a tendency not to provide medication intervention. Although ductus arteriosus quickly closes itself after birth in normal term infants, however, the dynamic changes detail of ductus arteriosus in preterm infants are unknown.

ELIGIBILITY:
Inclusion Criteria:

* less than 32 weeks' gestational age
* admission with 1 hours after birth

Exclusion Criteria:

* congenital abnormalities
* parents' refusal

Ages: 1 Minute to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: very preterm infants and extremely preterm infants with respiratory distress syndrome (RDS) and without RDS were included.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of patent ductus arteriosus(PDA) | three months after birth
  when did the ductus arteriosus close
dynamic changes of ductus arteriosus in diameter, velocity and direction of blood flow | after admission, 12 hour, 24 hour, 48 hour, 72 hour, 96 hour, 120 hour, 144 hour, 168 hour, 192 hour, 216 hour, 240 hour and 2 weeks or any time of ductus arteriosus closed
  dynamic changes of ductus arteriosus in diameter, velocity and direction of blood flow were measured

SECONDARY OUTCOMES:
the incidence of bronchopulmonary dysplasia | 36 weeks' gestational age
  whether or not bronchopulmonary dysplasia was assessed in 36 weeks' gestational age
the incidence of intraventricular hemorrhage(IVH) | 36 weeks' gestational age
  whether or not intraventricular hemorrhage(IVH) was assessed
necrotizing enterocolotis(NEC) | 36 weeks' gestational age
  whether or not NEC was assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Children's hospital of Chonqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
after paper published
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after paper published
Access Criteria: Email to neurochenlong@126.com